CLINICAL TRIAL: NCT03135314
Title: The Effect of Cocoa Flavanol Intake on Cerebral and Muscle Perfusion and Oxygenation in Hypoxia - Implications for Cognitive and Exercise Performance
Brief Title: Cocoa Flavanol Intake and Exercise in Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Lieselot Decroix, Principal investigator at Human Physiology research group, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CFEH2016
Record Dates: First submitted 2017-04-19; First posted 2017-05-01 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Hypoxia, Altitude
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hypoxia Cocoa flavanol (Active Comparator): Exercise or cognitive test in (acute) hypoxic condition after 7 days of cocoa flavanol intake
  Interventions: Dietary Supplement: cocoa flavanol
- Hypoxia Placebo (Placebo Comparator): Exercise or cognitive test in (acute) hypoxic condition after 7 days of placebo intake
  Interventions: Dietary Supplement: placebo
- Normoxia Cocoa flavanol (Active Comparator): Exercise or cognitive test in normoxic condition after 7 days of cocoa flavanol intake
  Interventions: Dietary Supplement: cocoa flavanol
- normoxia placebo (Placebo Comparator): Exercise or cognitive test in normoxic condition after 7 days of placebo intake
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: cocoa flavanol — 7 days intake of cocoa flavanol supplement (naturex)
  Arms: Hypoxia Cocoa flavanol; Normoxia Cocoa flavanol
Dietary Supplement: placebo — 7 days of placebo intake
  Arms: Hypoxia Placebo; normoxia placebo

SUMMARY:
Not uncommonly, sports events take place or finish at high altitude, where physical and cognitive (e.g. decision-making, motor control) performance in hypoxia is determining the outcome of sports performance. With nutritional supplements growing in popularity in the athletic and non-athletic population, research is increasingly focussing on dietary constituents which can improve cognitive and exercise performance.

Flavonoids, a subgroup of polyphenols, are a class of natural compounds found in the human diet and include subcategories of flavanols, flavonols, iso-flavones, flavones, and anthocyanidins. Intake of flavanols, found in grapes, tea, red wine, apples and especially cocoa, causes an nitric oxide (NO)-mediated vasodilatation and can improve peripheral and cerebral blood flow (CBF).

For cocoa flavanol (CF), there is evidence that both long term and acute intake can improve cognitive function, with the quantity and bioavailability of the consumed CF highly influencing its beneficial effects and with higher doses eliciting greater effects on cognition. Increased CBF following acute and chronic (3 months) CF intake has been demonstrated in healthy young subjects. Moreover, cognitive performance and mood during sustained mental efforts are improved after acute CF intake in healthy subjects and CF intake can increase prefrontal oxygenation during cognitive tasks in well-trained athletes. Moreover, CF intake is not only associated with an improved blood flow, but it might also improve exercise performance following 2 weeks of dark chocolate intake. On top of that, CF is known to have anti-oxidant properties and 2 week CF intake has been associated with reduced oxidative-stress markers following exercise.

In hypoxic conditions, arterial pressure of oxygen (PaO2) and arterial saturation of O2 (SaO2) are decreased, compromising tissue oxygen delivery. Since brain function and brain integrity are dependent on continuous oxygen supply, brain desaturation may result in an impaired cognitive function in hypoxia. The severity of the impairment is related to the extent of high altitude, with at 3000m (=14.3 % oxygen (O2); = 71% of oxygen available at sea level) psychomotor impairments being visible. Cerebral oxygenation, which can be measured by Near-infrared spectroscopy, is lowered in hypoxia.

It remains unclear whether CF intake can influence cerebral oxygenation and perfusion in hypoxic conditions and whether CF intake could (partially) counteract hypoxia-induced cognitive impairments. Therefore, the first aim of this study was to investigate whether cognitive function and prefrontal oxygenation during a mental demanding task will be impaired by hypoxic conditions (3000m altitude; 14.3% O2) and whether these impairments can be partially restored by subchronic CF intake (7 days, 900 mg/day).

Hypoxia also impairs physical performance. Hypoxia-induced reductions in cerebral oxygenation may favour central fatigue, i.e. the failure of the central nervous system to excite the motoneurons adequately, hence impairing exercise performance in hypoxic conditions. Since hypoxia also impairs oxygen delivery to muscle tissue, the decreased oxygen supply to and impaired oxidative energy production in the exercising muscle is a second factor negatively affecting exercise performance.

Besides the aforementioned effects of altitude on O2 delivery, hypoxia also results in increased oxidative stress. Oxidative stress refers to the imbalance between prooxidant and antioxidant levels in favor of prooxidants in cells and tissues and can result from diminished antioxidant levels or increased production of reactive oxygen species. The latter can be induced by both exhaustive exercise and high altitude. Since oxidative stress can be counteracted by CF, we also aim to investigate how markers of oxidative stress can be affected by CF intake by exercise in hypoxia. Therefore, the second aim of this study was to investigate possible beneficial effects of CF intake on changes in cerebral and muscle vasoreactivity and oxidative stress during exercise in hypoxia and its implications on exercise performance.

ELIGIBILITY:
Inclusion Criteria:

* train more than 10 hours/week

Exclusion Criteria:

* severe head injuries in the past
* hypertensive
* with cardiovascular disease / take medication for cardiovascular disease
* smokers
* take nutritional supplements
* had stayed at high altitude (>3000m) for 3 weeks during the last 6 months

Ages: 18 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
prefrontal/muscular oxygenation | change from baseline (pre-exercise) at post-exercise after 7 days of intake
work (kj) performed during 20 minute time trial | after 7 days of intake

SECONDARY OUTCOMES:
Flow mediated dilation | after 6 days of intake
oxidative stress | change from baseline (pre-exercise) at post-exercise after 7 days of intake

REFERENCES:
- [Derived] Decroix L, Tonoli C, Lespagnol E, Balestra C, Descat A, Drittij-Reijnders MJ, Blackwell JR, Stahl W, Jones AM, Weseler AR, Bast A, Meeusen R, Heyman E. One-week cocoa flavanol intake increases prefrontal cortex oxygenation at rest and during moderate-intensity exercise in normoxia and hypoxia. J Appl Physiol (1985). 2018 Jul 1;125(1):8-18. doi: 10.1152/japplphysiol.00055.2018. Epub 2018 Mar 15. PMID 29543135